CLINICAL TRIAL: NCT07095647
Title: Surgical Outcomes of Simultaneous Hysteroscopy/Laparoscopy for Cesarean-Section Niche Ectopic Pregnancy Management and Uterine Niche Repair
Brief Title: Surgical Management of Cesarean Scar Ectopic Pregnancy: Hysteroscopy & Laparoscopy Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Shereen Naguib, Lecturer of Obstetrics & Gynecology, Faculty of Medicine, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC 9.6.2025
Record Dates: First submitted 2025-07-30; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — Hysteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cesarean Scar Ectopic Pregnancy Patients (CSEP) (Other): Patients presenting pregnant with a history of at least one previous Cesarean Section, and Transvaginal ultrasound documentation of Cesarean Scar Ectopic Pregnancy.
  Interventions: Procedure: Hysteroscopy

INTERVENTIONS:
Procedure: Hysteroscopy — Hysteroscopic-guided suction evacuation and double-layer laparoscopic repair of the niche were performed concomitantly and followed by second-look hysteroscopy to ensure the competence of the repair.

SUMMARY:
The study investigates the feasibility, safety, and outcomes of a simultaneous surgical approach for cesarean scar ectopic pregnancy (CSEP). CSEP is a prevalent and serious form of ectopic pregnancy requiring swift intervention. The research explores using hysteroscopy and laparoscopy concurrently to manage the CSEP and repair the uterine scar defect. The procedure involved hysteroscopic-guided evacuation and a double-layer laparoscopic repair, followed by a second hysteroscopy to confirm the repair's effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients with positive clinical and lab pregnancy diagnosis;
* Patients with history of at least one previous Cesarean section;
* Patients with Transvaginal ultrasound documenting Cesarean scar ectopic Pregnancy;

Exclusion Criteria:

* Patients with were extensive adhesions between the mass and the urinary bladder on MRI;
* Patients with myomas, polyps, endometrial hyperplasia, and cancers of the cervix or endometrium;
* Patients with a body mass index (BMI) of >35kg/m2;
* Patients with previous abdominal surgeries with possible difficulties during laparoscopy;
* Patients with menstrual irregularities, or coagulation disorders.

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Success Rate of Hysteroscopy in Restoring the normal endometrial metrics, and removing any uterine defects. | 6~7 months
  The proportion of patients who restored their normal endometrial metrics and removed any uterine scars during the study, reflecting the effectiveness of the applied Hystreoscopy regimens.

CONTACTS AND LOCATIONS:
Locations (1):
- Banha University, Banhā, El- Qalyobia, Egypt